CLINICAL TRIAL: NCT06387862
Title: Pharmacokinetics of Inhaled Levosimendan
Acronym: Symbiov
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2022SIMBIOV
Record Dates: First submitted 2024-01-09; First posted 2024-04-29 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2023-10

CONDITIONS: Left Ventricular Dysfunction
Keywords: levosimendan; inhalation; pharmakokinetic
MeSH Terms: conditions — Ventricular Dysfunction, Left; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levosimendan inhalation (Experimental): Levosimendan 12µg/kg inhalation over 10 minutes, once
  Interventions: Drug: Levosimendan 2.5 milligram/milliliter Injectable Solutiondose Inhaled
- Levosimendan intravenous (Active Comparator): Levosimendan 12µg/kg intravenous over 10 minutes, once
  Interventions: Drug: Levosimendan 2.5 milligram/milliliter Injectable Solutiondose Intravenous

INTERVENTIONS:
Drug: Levosimendan 2.5 milligram/milliliter Injectable Solutiondose Inhaled — Each patient will receive 12µg/kg of levosimendan by inhalation over 10 min. During 10h following inhaled dose, plasma concentrations will be measured.
  Arms: Levosimendan inhalation
Drug: Levosimendan 2.5 milligram/milliliter Injectable Solutiondose Intravenous — Each patient will receive 12µg/kg of levosimendan by intravenous (IV) administration over 10 min and at the same timepoints plasma samples will be measured
  Arms: Levosimendan intravenous

SUMMARY:
Determination of biological availability, time-to-peak and elimination half-life of inhaled levosimendan by administration of an inhaled- and intravenous dose of levosimendan.

ELIGIBILITY:
Inclusion Criteria:

* Subject >18 years of age
* Scheduled for elective coronary artery bypass grafting (CABG)
* Provided written informed consent
* Impaired left ventricular function (LVEF <40%)

Exclusion Criteria:

* Known allergy for levosimendan or solutes
* Persistent angina, defined as Canadian Cardiovascular Society score > I
* History of valvular intervention or uncorrected primary stenotic valve disease
* Uncorrected thyroid disease
* Infiltrative, hypertrophic or restrictive cardiomyopathy
* Pericardial disease
* Active myocarditis
* Chronic obstructive pulmonary disease requiring long-term treatment with β-agonists, Theophylline, or corticosteroids (FEV1 < 80%; Tiffeneau-index <0.7)
* History of serious arrhythmias, defined as a history of ventricular tachycardia or fibrillation other than that occurring within 24 hours after acute myocardial infarction (MI)
* resting heart rate > 115 bpm for at least 10 minutes on repeated measurements
* Supine systolic blood pressure < 85 mm Hg or >200 mm Hg
* patients with implanted pacemaker/defibrillator or cardiac resynchronisation therapy (CRT-device)
* primary renal or hepatic impairment (creatinine > 2.5 mg/dL or aspartate aminotransferase/alanine aminotransferase >2 times upper limit of normal and/or increased level of bilirubin (> 2 times the upper limit of normal and increase of international normalised ratio (INR) above the upper limit of normal, respectively)
* Uncorrected hypokalemia or hyperkalemia (potassium <3.5 mmol/L or >5.5 mmol/L)
* Uncorrected hypomagnesemia (magnesium <0.65mmol/L)
* Treatment with another investigational agent within 30 days before study entry
* Intubated and mechanically ventilated at the time of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Bioavailability of inhaled levosimendan | Baseline, plasma samples at 5 minutes, 10 minutes, 15 minutes, 20 minutes, 30 minutes, 45 minutes, 1 hour, 1hour 30 minutes, 2 hours , 3 hours , 6 hours, 10 hours after end of infusion/inhalation
  Assessment of bioavailability of inhaled levosimendan in spontaneous breathing patients,
Time-to-peak of inhaled levosimendan | Baseline, plasma samples at 5 minutes, 10 minutes, 15 minutes, 20 minutes, 30 minutes, 45 minutes, 1 hour, 1hour 30 minutes, 2 hours , 3 hours , 6 hours, 10 hours after end of infusion/inhalation
  Assessment of time-to-peak plasma concentration of inhaled levosimendan in spontaneous breathing patients
Elimination half-life of inhaled levosimenan | Baseline, plasma samples at 5 minutes, 10 minutes, 15 minutes, 20 minutes, 30 minutes, 45 minutes, 1 hour, 1hour 30 minutes, 2 hours , 3 hours , 6 hours, 10 hours after end of infusion/inhalation
  Assessment of elimination half-life of inhaled levosimendan in spontaneous breathing patients

SECONDARY OUTCOMES:
Effect of inhaled levosimendan on MAP | Baseline, plasma samples at 5 minutes, 10 minutes, 15 minutes, 20 minutes, 30 minutes, 45 minutes, 1 hour, 1hour 30 minutes, 2 hours , 3 hours , 6 hours, 10 hours after end of infusion/inhalation
  Assessment of effect of inhaled levosimendan on invasively-measured hemodynamic parameter mean arterial blood pressure (MAP)
Effect of inhaled levosimendan on TVR | Baseline, plasma samples at 5 minutes, 10 minutes, 15 minutes, 20 minutes, 30 minutes, 45 minutes, 1 hour, 1hour 30 minutes, 2 hours , 3 hours , 6 hours, 10 hours after end of infusion/inhalation
  Assessment of effect of inhaled levosimendan on invasively-measured hemodynamic parameter total vascular resistance (TVR)
Effect of inhaled levosimendan on CO | Baseline, plasma samples at 5 minutes, 10 minutes, 15 minutes, 20 minutes, 30 minutes, 45 minutes, 1 hour, 1hour 30 minutes, 2 hours , 3 hours , 6 hours, 10 hours after end of infusion/inhalation
  Assessment of effect of inhaled levosimendan on invasively-measured hemodynamic parameter Cardiac Output (CO)
Effect of inhaled levosimendan on LVOT VTI | Baseline, plasma samples at 5 minutes, 10 minutes, 15 minutes, 20 minutes, 30 minutes, 45 minutes, 1 hour, 1hour 30 minutes, 2 hours , 3 hours , 6 hours, 10 hours after end of infusion/inhalation
  Assessment of effect of inhaled levosimendan on echocardiography-derived parameter left -ventricular-outflow-tract (LVOT) velocity-time-integral (VTI) as marker for cardiac output
Effect of inhaled levosimendan on FAC of the right vetricle | Baseline, plasma samples at 5 minutes, 10 minutes, 15 minutes, 20 minutes, 30 minutes, 45 minutes, 1 hour, 1hour 30 minutes, 2 hours , 3 hours , 6 hours, 10 hours after end of infusion/inhalation
  Assessment of effect of inhaled levosimendan on echocardiography-derived parameter Fractional-Area-Change (FAC) of the right ventricle as marker of right ventricular function
Effect of inhaled levosimendan on S' | Baseline, plasma samples at 5 minutes, 10 minutes, 15 minutes, 20 minutes, 30 minutes, 45 minutes, 1 hour, 1hour 30 minutes, 2 hours , 3 hours , 6 hours, 10 hours after end of infusion/inhalation
  Assessment of effect of inhaled levosimendan on echocardiography-derived parameter S' wave velocity as marker of right ventricular function
Effect of inhaled levosimendan on SPAP | Baseline, plasma samples at 5 minutes, 10 minutes, 15 minutes, 20 minutes, 30 minutes, 45 minutes, 1 hour, 1hour 30 minutes, 2 hours , 3 hours , 6 hours, 10 hours after end of infusion/inhalation
  Assessment of effect of inhaled levosimendan on echocardiography-derived parameter (SPAP) systolic pulmonary artery pressure

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Raes, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No